CLINICAL TRIAL: NCT00247884
Title: Directly Observed Therapy for the Treatment of Hepatitis C Virus Infection in Injection Drug Users
Brief Title: Pender Assisted Therapy (PATh) - Prospective Study of the Treatment of HCV
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Brian Conway, University of British Columbia
Other Study IDs: C05-0219
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Hepatitis C Virus Infection
Keywords: Injection drug users; pegylated interferon; ribavirin,; HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The treatment of HCV-infected IDUs presents multiple challenges, such as adherence to therapy, relapse of substance use, re-infection, and co-morbid psychiatric disease. Some guidelines recommended that IDUs not be offered HCV treatment until they had stopped all such use for > 6 months, raising some questions about fairness and discrimination. Little published data exist on HCV therapy in active IDUs. However, extensive evidence exists that, when specific programs are developed, IDUs can be successfully engaged in care. In IDUs, strategies shown to improve adherence include directly-observed therapy (DOT), cash incentives, and comprehensive case management. Weekly interferon dosing now provides a means of improving HCV treatment adherence, and makes a DOT approach more practical. Within an observational, prospective clinical cohort, we will be able to identify a group of IDUs infected with HCV genotype 2 or 3 who would most benefit from treatment for their infection. We will design a systematic approach to the determination of their appropriateness for treatment, refine the approach to their treatment within a directly observed therapy (DOT) setting, and evaluate the success of the approach (defined as the achievement of Sustained Virologic Response (SVR)). Taken together, this project will help define a systematic approach to HCV infection in the inner city. The hypothesis is that the development of a systematic approach for the diagnosis of HCV and the establishment of a directly observed therapy (DOT) program for the treatment of HCV infection in IDUs will constitute an effective means of controlling the epidemic of this infection within this population.

DETAILED DESCRIPTION:
We will evaluate up to 200 IDUs receiving care in our clinics. For those found to carry genotype 2 or 3 and be eligible for treatment on medical grounds, we will evaluate the patients in a bi-weekly case conference. All physicians who are participating in this study will also be included. Nursing and counselling staff will also be present. For those who qualify to receive therapy for HCV, based on Provincial guidelines, a decision will be made regarding their appropriateness to begin treatment based on physical, mental, social and addiction-related factors. Once treatment is initiated, the primary objective of this study is to evaluate a relatively high intensity DOT program for the treatment of HCV-infected IDUs. All patients will have access to: full-time primary care physician, half-time specialist physician, immediate access to one of three full-time nurses and one of six full-time counsellors. All weekly pegylated interferon injections and one of two daily doses of oral medications will be administered/witnessed by clinic staff. The interferon will be injected at the clinic by a staff nurse, while the one daily dose of ribavirin that will be observed will be given simultaneously with methadone (if the patient is on maintenance therapy with this agent) either at the clinic site or at a community pharmacy, as has been decided in that individual's plan of care. This plan will be maintained at the time of initiation of HCV therapy. This study will evaluate 50 individuals infected with HCV genotypes 2/3 receiving up to 24 weeks of therapy. The primary outcome will be evaluation of SVR (undetectable virus at 48 weeks, 24 weeks after cessation of therapy). Patients will be enrolled at PCHC, TPHU or CCHC, according to their usual site of medical care. They will be assessed to determine if they wish to participate in the trial and meet its inclusion and exclusion criteria. They will then be asked to provide written, informed consent using the document approved by the Research Ethics Board. Once consent is granted, a medical evaluation and laboratory testing will be completed. Clinical data will consist of a medical history (to include recreational drug use history) and physical examination (to include vital signs, weight and height). Laboratory evaluations will include: confirmation of HCV antibody status, viremia and genotype; Hematology (CBC); Blood Chemistry (ALT, creatinine, alkaline phosphatase, total bilirubin (direct and indirect), urea nitrogen, albumin, glucose, sodium, potassium, chloride); ANA, TSH, HBsAg, iron studies, ceruloplasmin, AFP, PT/INR, HIV antibody test (CD4 cell count and HIV plasma viral load, if known HIV-positive); Urinalysis and Toxicology Screen; Serum pregnancy test in women of child-bearing potential. All blood work to evaluate treatment efficacy and toxicity will be collected by study personnel. This will be done at weeks 2, 4, 6, 8, 12, 16, 20 and 24 (more frequently if clinically indicated), according to the standard of care. All medical follow-up will be according to standard of care. This study will involve the prospective evaluation of HCV therapy in patients who would receive treatment regardless of their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

Age greater than 18 years; Serum HCV-RNA positive; HCV genotype 2 or 3; HBsAg negative; serum ALT greater than 1.5x upper limit normal greater than 3 months; Agreement from each participant of childbearing age to practice contraception; Ability to provide informed consent; judged to be appropriate for immediate treatment by case conference.

Exclusion Criteria:

Any cause for chronic liver disease other than HCV (including alcohol use greater than 350 g/wk); Pregnant or breastfeeding women; Active HBV infection; Hemolytic anemia; Decompensated cirrhosis or portal hypertension; Active suicidal ideation, psychosis, mania or hypomania; Serum creatinine greater than 180 µg/mL; Hemoglobin less than 120 g/L in men or 110 g/L in women; Platelets < 90 x 109/L; Neutrophils less than 1.5 x 109/L; Active autoimmune disease; NYHA disease > grade 2; Psoriasis requiring systemic therapy; Active malignancy apart from non melanoma skin cancer; Use of systemic immunosuppressant agents; Weight greater than 105 kg ; Prior treatment of HCV with interferon or ribavirin; HIV positive with CD4 count less than 250 cells/mm3 or receiving didanosine (due to interaction with ribavirin); Life expectancy less than 2 years; judged to be inappropriate for immediate treatment by case conference

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Injection drug users
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2005-06; Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Conway, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Pender Community Health Centre, Vancouver, British Columbia
  - Cool-Aid Community Health Centre, Victoria, British Columbia